CLINICAL TRIAL: NCT07405606
Title: Psilocybin-assisted Therapy for Comorbid Major Depressive Disorder and Alcohol Use Disorder: A Pilot Randomized Clinical Trial
Brief Title: Psilocybin-assisted Therapy for Comorbid Major Depressive Disorder and Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 071/2023
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD); Alcohol Use Disorder (AUD)
Keywords: depression; psilocybin; alcohol use disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism; Depression | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin (25 mg) (Experimental): Participant is administered one oral capsule (25 mg psilocybin) with water.
  Interventions: Drug: Psilocybin 25 mg
- Placebo (Placebo Comparator): Participant is administered one oral capsule (0 mg psilocybin) with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin 25 mg — Participants will orally consume Psilocybin (25 mg) with water.
  Arms: Psilocybin (25 mg)
Drug: Placebo — Participants will orally consume placebo matching the intervention with water.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the safety and efficacy of psilocybin assisted Therapy (PAT) in individuals with comorbid Major Depressive Disorder (MDD) and Alcohol Use Disorder (AUD). The main question it aims to answer is:

- What is the feasibility and safety of administering PAT in adults with MDD-AUD by evaluating recruitment, retention, tolerability, and safety?

Researchers will compare the psilocybin (25 mg) and placebo groups to see if there are any significant differences in frequency of dropouts or serious adverse events.

Participants will:

* be randomized to receive either psilocybin (25 mg) or placebo
* visit the site (in-person and remotely) for a total of 14 times to complete study tasks
* receive psilocybin-assisted therapy (PAT) at five various timepoints

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Must be deemed to have capacity to provide informed consent;
* Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent;
* Stated willingness to comply with all study procedures;
* Be deemed in health compatible with the study procedures according to study physician;
* Ability to take oral medication and be willing to adhere to the PAT regimen;
* Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation;
* Fulfil Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5) criteria for a primary diagnosis of current single or recurrent episodes of MDD of at least moderate severity but without psychotic features and a comorbid AUD diagnosis (moderate or severe) using the SCID-5;
* A score of at least 14 on the Hamilton Depression Rating Scale for Depression (HAMD);
* Participants should not be interested in initiating standard pharmacotherapies for MDD or AUD. The need to start/resume standard pharmacotherapies will be reassessed at Week 6.
* Individuals who are willing to and tapered off current antidepressant or IMAOs, antipsychotic and anti-alcohol/anti-craving medications for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose physician confirms that it is safe for them to do so;
* Individuals who are willing to and have tapered off current inhibitors of 5'-diphospho-glucuronosyltransferase (UGT)1A9 and 1A10, aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs) for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose physician confirms that it is safe for them to do so;
* Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

* Pregnant as assessed by a urine pregnancy test at Screening (V1) and Baseline (V2) or individual's that intend to become pregnant during the study or are breastfeeding;
* Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension (over 160/100 mmHG), low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment.
* Diagnosis of cirrhosis, AST or ALT elevations > 3x upper limit of normal; significant abnormal liver function that would preclude administration of psilocybin based on the judgement of the QI (assessed notably by bilirubin, albumin, alkaline phosphatase, GGT, and INR functions)
* Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder; obsessive-compulsive disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the SCID-5 clinical interview;
* Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder as determined by the family medical history form and discussions with the participant;
* Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) score > 9, or any other indication that the participant may experience medically complicated withdrawal from alcohol, such as a score of ≥4 in the Prediction of Alcohol Withdrawal Severity Scale.
* Use benzodiazepines (with the exception of use of up to 2mg of lorazepam equivalent per day for insomnia and anxiety if it is not taken within 12 hours before the psilocybin dose (Week 2).
* Have a DSM-5 diagnosis of substance use disorder (excluding alcohol, cannabis, tobacco and caffeine) within the preceding 6 months;
* Presence of baseline prolonged QTc (more than 0.45 seconds for males and 0.47 seconds for females) or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors;
* Use of aldehyde dehydrogenase (ALDH) inhibitors and UDG modulators;
* Use of hallucinogens in the past 5 years; or total hallucinogen use ≥10 times)
* Current suicidality risk as indicated during the conduct of the Columbia Suicide Severity Rating Scale (C-SSRS) with concurrence after a study physician's evaluation if the response to C-SSRS questions 1 or 2 is "yes")
* Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.
* Participants that are responding to anti-alcohol or anti-craving medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Adherence | Week 2 (Visit 4)
  Although all administration of psilocybin will be administered by qualified staff, the investigators will measure adherence through visit compliance (i.e., missed visits).
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess changes in depressive symptoms on a 10-item scale with each item rated on a scale of 0-6. Higher scores indicate greater severity of symptoms.
Hamilton Depression Rating Scale (HAMD-17) | 4-week post dose; week 26.
  Used to assess changes in depressive symptoms using 3-point (0-2) or 5-point (0-4) Likert scales. Higher scores indicate greater severity of symptoms.
Quick Inventory of Depressive Symptomatology - Self Report (QUIDS-SR) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess changes in depressive symptoms with a minimum score of 0 to a maximum score of 27.
Alcohol Timeline Followback (TLFB) | Baseline; week 2 (visit 3); 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  To monitor alcohol consumption, heavy drinking days, drinks per day, drinks per drinking day, percent very heavy drinking days, percent participants with no heavy drinking days, and abstinent percent will be measured.
Clinical Institute Withdrawal Assessment (CIWA) | Baseline; week 2 (visit 3); week 2 (visit 4); 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess alcohol withdrawal symptoms. Scores range from 0 to 67 with higher scores indicating greater severity of withdrawal symptoms.
Prediction of Alcohol Withdrawal Severity Scale (PAWSS) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess risk of alcohol withdrawal symptoms using a 10-item scale with the total score ranging from 0 to 10. Higher scores indicate greater risk of withdrawal symptoms.
Penn Alcohol Craving Scale (PACS) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess history, frequency, and consequences of alcohol use. Scores range from 0 to 30 with higher scores indicating greater craving.
Addiction Severity Index (ASI) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post dose; 4-week post dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess history, frequency, and consequences of alcohol use

SECONDARY OUTCOMES:
5 Dimensional Altered States of Consciousness (5-DASC) | Week 2 (visit 4).
  Used to assess subjective effects of psilocybin.
Psychological Insight Questionnaire (PIQ) | Week 2 (visit 4).
  Used to assess subjective effects of psilocybin. Contains 23 items rated on a 5-point Likert scale.
Mystical Experience Questionnaire (MEQ) | Week 2 (visit 4).
  Used to assess subjective effects of psilocybin. Contains 30 items rated on a 5-point Likert scale.
Challenging Experience Questionnaire (CEQ) | Week 2 (visit 4).
  Used to assess subjective effects of psilocybin. Contains 26 items rated on a 5-point Likert scale.
General Anxiety Disorder-7th edition (GAD-7) | Baseline; week 26.
  Used to assess anxiety-related symptoms. Scores range from 0 to 21 with higher scores indicating greater severity of anxiety symptoms.
State Trait Anxiety Index (STAI) | Baseline; week 26.
  Used to assess anxiety-related symptoms. Scores range from 20 to 80 with higher scores indicating greater severity of anxiety symptoms.
World Health Organization Quality of Life Questionnaire Brief Version (WHOQOL-BREF) | Baseline; week 26.
  Used to assess overall quality of life. Scores range from 0 to 100 with higher scores indicating greater quality of life.
Big Five Inventory (BFI) | Baseline; week 26.
  Used to assess personality. Contains 44 items with each item rated on a five-point Likert scale from 1 (disagree a lot) to 5 (agree a lot). Higher scores in each trait indicates stronger association to the trait.
Pittsburgh Sleep Quality Index (PSQI) | Baseline; week 26.
  Used to assess quality of sleep. Score ranges from 0 to 21 with higher scores indicating greater disturbance to sleep.
Acceptance & Action Questionnaire II (AAQ-II) | Baseline; 1-day post dose; 1-week post dose; 2-week post dose; 3-week post-dose; 4-week post-dose; week 10; week 14; week 18; week 22; week 26.
  Used to assess psychological flexibility. There are 7-items each rated on a 7-point Likert scale. Higher scores indicate greater psychological inflexibility.
Stanford Expectations of Treatment Scale (SETS) | Baseline
  Used to assess participants' positive and negative treatment expectancies.
Working Alliance Inventory (WAI) | Week 2 (visit 3); 1-day post dose; 1-week post dose.
  Used to assess the participants' therapeutic relationship with their therapists. Scores range from 12 to 60 with higher scores indicating stronger therapeutic alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No